CLINICAL TRIAL: NCT00383019
Title: A 8-WEEK, RANDOMIZED, DOUBLE-MASKED, PARALLEL GROUP, PHASE III STUDY COMPARING THE EFFICACY AND SAFETY OF XALACOM AND XALATAN IN PATIENTS WITH PRIMARY OPEN ANGLE GLAUCOMA (POAG) OR OCULAR HYPERTENSION (OH)
Brief Title: A Study Comparing Xalacom And Xalatan In Patients With Primary Open Angle Glaucoma (POAG) Or Ocular Hypertension (OH).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6641050
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Xalacom

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Xalatan (Experimental)
  Interventions: Drug: Xalatan
- Xalacom (Experimental)
  Interventions: Drug: Xalacom

INTERVENTIONS:
Drug: Xalatan — latanoprost 0.005%, one rop once daily in evening
  Arms: Xalatan
Drug: Xalacom — latanoprost 0.005% adn timolol 0.5%, one drop, once daily
  Arms: Xalacom

SUMMARY:
This study will examine the efficacy and safety of Xalacom comparing with those of Xalatan in Japanese patients with POAG or OH, in order to show superiority of Xalacom over Xalatan in efficacy and similarity of safety between Xalacom and Xalatan.

ELIGIBILITY:
Inclusion Criteria:

* Intraocular pressure is 18 mmHg or more at baseline after treatment with Xalatan for 4 weeks or more.

Exclusion Criteria:

* History of no-response to timolol
* History of trabeculectomy
* History of other ocular surgery including ALT, SLT,and trabeculotomy within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-11-14 (Actual); Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- Japan (54):
  - Nomura Eye Clinic, Ichinomiya, Aichi-ken
  - Matsusura Eye Clinic, Ichinomiya, Aichi-ken
  - Yasuma Eye Clinic, Nagoya, Aichi-ken
  - TANABE Eye Clinic, Nagoya, Aichi-ken
  - Suzuki Eye Clinic, Nagoya, Aichi-ken
  - Mitsuhashi Eye Clinic, Narashino, Chiba
  - Ohtsuka Eye Clinic, Sapporo, Hokkaido
  - Sasamoto Eye Clinic, Sapporo, Hokkaido
  - Ohyachi Kyouritsu Eye Clinic, Sapporo, Hokkaido
  - Kaimeido Eye Clinic, Sapporo, Hokkaido
  - Kobe University Hospital, Koube, Hyōgo
  - Kanazawa university hospital, Kanazawa, Ishikawa-ken
  - Lumine Hatano Eye Clinic, Fujisawa, Kanagawa
  - Tanino clinic, Kamakura, Kanagawa
  - Aoki eye clinic, Sagamihara, Kanagawa
  - Kikuna Yuda Eye Clinic, Yokohama, Kanagawa
  - Fujita Eye Clinic, Sapporo, Kokkaido
  - Chihara Eye Clinic, Uji, Kyoto
  - Miyata Eye Hospital, Miyakonojō, Miyazaki
  - Hayashi Eye Clinic, Kumagaya, Saitama
  - Hiraoka Eye Clinic, Tokorozawa, Saitama
  - Hanasaki Eye Clinic, Fuji, Shizuoka
  - Nakajima Eye Clinic, Fuji, Shizuoka
  - Yoshimura Eye & Internal Medical Clinic, Mishima, Shizuoka
  - Muramatsu Ganka Clinic, Susono, Shizuoka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Police Hospital, Chiyoda City, Tokyo
  - Ochanomizu Inoue Eye Clinic, Chiyoda-ku, Tokyo
  - Keio Hachioji Matsumoto Eye Clinic, Hachiōji, Tokyo
  - Manabe Clinic, Hamura, Tokyo
  - Tokyo Sugita Eye Center, Katsushika-ku, Tokyo
  - Kiyosenomori Hospital, Kiyose, Tokyo
  - Miyazaki Eye Clinic, Koto-ku, Tokyo
  - Takase Ganka Tairamachi Clinic, Meguro City, Tokyo
  - Ohashi Eye Clinic, Meguro-ku, Tokyo
  - Kunitoshi Eye Clinic, Musashino, Tokyo
  - Shimizu Eye Clinic, Musashino, Tokyo
  - WAKABA Eye Clinic, Ōta-ku, Tokyo
  - Seijo Clinic, Setagaya City, Tokyo
  - Yotsuya Shirato Ganka, Shinjuku, Tokyo
  - Tachihi Bill clinic, Tachikawa, Tokyo
  - Ueno Eye Clinic, Taito-ku, Tokyo
  - Hayashi Eye Hospital, Fujuoka
  - Hayashi Tennjin Eye Clinic, Fukuoka
  - Ohshima Hospital of Opthalmology, Fukuoka
  - Kato Eye Clinic, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Niigata University Medical and Dental Hospital, Niigata
  - Nishi Eye Hospital, Osaka
  - Adachi Eye Clinic, Osaka
  - Osaka Welfare Pension Hospital, Osaka
  - Nanba Opthalmology, Shizuoka
  - Sugita Eye Hospital, Sugita

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641050&StudyName=A%20Study%20Comparing%20Xalacom%20And%20Xalatan%20In%20Patients%20With%20Primary%20Open%20Angle%20Glaucoma%20%28POAG%29%20Or%20Ocular%20Hypertension%20%28OH%29.%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 centers in Japan
Pre-assignment Details: 300 subjects were treated with Xalatan in Run-in period. (Run-in period: subjects treated with Xalatan(0.005% latanoprost eye drop), one drop, once daily in the evening (20:00-23:00).) Of these, 289 subjects were assigned to groups (144 in KP2035 group and 145 in Xalatan group).
Groups:
- KP2035 Group: Subjects were treated with KP2035 (0.005% latanoprost + 0.5% timolol combination eye drop) one drop, once daily in the evening (20:00-23:00).
- Xalatan Group: Subjects were treated with Xalatan (0.005% latanoprost), one drop, once daily in the evening (20:00-23:00).
Period: Overall Study
Arm/Group | KP2035 Group | Xalatan Group
Started | 144 | 145
Completed | 139 | 143
Not Completed | 5 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KP2035 Group | Xalatan Group | Total
Number analyzed (Participants) | 144 | 145 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 77 | 155
  >=65 years | 66 | 68 | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 74 | 144
  Male | 74 | 71 | 145
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 144 | 145 | 289

OUTCOME MEASURES:

1. Primary Outcome: Change of Intraocular Pressure (IOP) From Baseline to Week 8
Description: Value at Week 8 minus value at baseline
Time Frame: Baseline to Week 8
Population: The primary efficacy analysis population was the Intent-to-treat population (ITT) which consisted of all subjects treated with the study drug as randomized. If there were any missing IOP values at Week 8, the data were supplemented by LOCF (Last Observation Carried Forward) using data at Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
mmHg | -2.59 [-2.92 to -2.25] | -1.62 [-1.96 to -1.28]

2. Secondary Outcome: Change of IOP From Baseline to Week 4
Description: Value at Week 4 minus value at baseline
Time Frame: Baseline to Week 4
Population: ITT
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
mmHg | -2.50 [-2.83 to -2.17] | -1.17 [-1.50 to -0.84]

3. Secondary Outcome: Number of Subjects With an IOP of <=15 mmHg at Week 8
Description: Number of subjects who achieved IOP reduction to 15 mmHg or below at Week 8
Time Frame: Week 8
Population: The efficacy analysis population was ITT. If there were any missing IOP values at Week 8, the data were supplemented by LOCF using data at Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 36 | 13

4. Secondary Outcome: Number of Subjects With an IOP of <=16 mmHg at Week 8
Description: Number of subjects who achieved IOP reduction to 16 mmHg or below at Week 8
Time Frame: Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 60 | 35

5. Secondary Outcome: Percent Change of IOP From Baseline to Week 8
Description: Value at Week 8 minus value at baseline was divided by baseline value, then multiplied by 100
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
percent change | -12.67 [-14.40 to -10.93] | -7.69 [-9.42 to -5.95]

6. Secondary Outcome: Number of Subjects With an IOP of <=18 mmHg at Week 8
Description: Number of subjects who achieved IOP reduction to 18 mmHg or below at Week 8
Time Frame: Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 105 | 91

7. Secondary Outcome: Number of Subjects With an IOP Reduction of >=2 mmHg From Baseline to Week 8
Description: Number of subjects whose IOP were reduced by 2 mmHg or more at Week 8 from baseline
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 95 | 65

8. Secondary Outcome: Number of Subjects With an IOP Reduction of >=3 mmHg From Baseline to Week 8
Description: Number of subjects whose IOP were reduced by 3 mmHg or more at Week 8 from baseline
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 66 | 40

9. Secondary Outcome: Number of Subjects With an IOP of <=17 mmHg at Week 8
Description: Number of subjects who achieved IOP reduction to 17 mmHg or below at Week 8
Time Frame: Week 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | KP2035 Group | Xalatan Group
Number analyzed (Participants) | 144 | 145
Participants | 83 | 60

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | KP2035 Group | Xalatan Group
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/145
Serious Adverse Events (participants affected / at risk) | 1/144 | 2/145
Other Adverse Events (participants affected / at risk) | 51/144 | 29/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KP2035 Group (N=144) | Xalatan Group (N=145)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KP2035 Group (N=144) | Xalatan Group (N=145)
Conjunctivitis (Eye disorders) | 2 | 1
Retinal tear (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 25 | 2
Nasopharyngitis (Infections and infestations) | 6 | 2
Tinea pedis (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 2 | 3
Pharyngitis (Infections and infestations) | 1 | 0
Glucose urine present (Investigations) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Punctate keratitis (Eye disorders) | 2 | 4
Eye pain (Eye disorders) | 0 | 2
Foreign body sensation in eye (Eye disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Meibomianitis (Eye disorders) | 0 | 1
Scleritis (Eye disorders) | 0 | 1
Growth of eyelashes (Eye disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.